CLINICAL TRIAL: NCT05648695
Title: Efficacy of Non-invasive NESA Neuromodulation in Fibromyalgia: a Randomised, Triple-blind Clinical Trial
Brief Title: Efficacy of Non-invasive NESA Neuromodulation in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NESA FIBRO
Record Dates: First submitted 2022-11-20; First posted 2022-12-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Fibromyalgia
Keywords: physical therapy modality; Pain; Chronic Fatigue Disorder; Sleep Quality
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue Syndrome, Chronic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive Neuromodulation (Experimental): Non-invasive Neuromodulation Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7 level.
  Interventions: Device: Non-invasive Neuromodulation
- Placebo Non-invasive Neuromodulation (Placebo Comparator): Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7.
  Interventions: Device: Placebo Non-invasive Neuromodulation

INTERVENTIONS:
Device: Non-invasive Neuromodulation — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, each session, until 13 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7. Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 millivolt and intensity 0.5 μA.
  Arms: Non-invasive Neuromodulation
Device: Placebo Non-invasive Neuromodulation — The same protocol described for the experimental group will be applied, but microcurrents device which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents.
  Arms: Placebo Non-invasive Neuromodulation

SUMMARY:
Fibromyalgia is a chronic condition that causes pain throughout the body, fatigue and other symptoms. Among the most common clinical symptoms are sleep and anxiety disorders. All these symptoms are very disabling and have a negative impact on the quality of life of these people.

There is currently no curative treatment for this pathology and current treatments focus their efforts on reducing the intensity of the symptoms. The current approach is mainly pharmacological, with the possible side effects that this entails.

DETAILED DESCRIPTION:
The NESA XSIGNAL® device is a non-invasive, low-frequency neuromodulation device that uses microcurrents to restore the electrical balance in the body. This technology is approved as medical equipment and is CE marked (attached in separate files).

This non-invasive neuromodulation equipment is beginning to show promising results in patients with sleep disorders. So it can be a useful tool to reduce the impact on the quality of life of people with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Diagnosis of Fibromyalgia meeting ACR 1990/20101,2 criteria, made by a physician, documented by a clinical report.
* Diagnosis of Fibromyalgia made at least 12 months ago
* Stable baseline treatment in the month prior to inclusion in the study
* Signed informed consent
* In normal condition and mentally competent to participate in the study.
* Able to complete the study questionnaires.

Exclusion Criteria:

* Have any of the following contraindications for treatment with NESA XSIGNAL®: pacemakers, internal bleeding, not applying electrodes to skin in poor condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and/or phobia of electricity.
* Failure to sign the informed consent form.
* Active chronic inflammatory joint diseases.
* Active neurological diseases with central or peripheral nervous system involvement.
* Active systemic autoimmune diseases
* Psychotic disorders
* Active concomitant neoplastic or infectious processes
* Medication changes in the month prior to study inclusion or throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Change in Pain assessed by VAS | Baseline and up to three weeks
  The instrument will be used to measure the change of pain before and after the intervention will be the Visual Analogue Scale (VAS).
  Participants will be asked to mark the level of their pain on a 100 mm, no hatched VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable".
Change in Sleep quality | Baseline and up to three weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used. It consists of 19 self-administered questions and 5 questions assessed by the patient's partner or roommate (if available). Only the self-administered questions are included in the score.
  The higher the total score, the worse the sleep quality. Thus, a total score less than or equal to five on the Pittsburgh scale indicates that, in general, your sleep quality is optimal, while a total score greater than five suggests that you have sleep problems, of greater or lesser severity.

SECONDARY OUTCOMES:
Functional capacity | Baseline and up to three weeks
  The fibromyalgia impact questionnaire (FIQ) will be used. It assesses the impact on health in terms of physical capacity, the ability to carry out usual work and, in the case of paid work, the degree to which fibromyalgia has affected this activity as well as subjective items closely related to this pathology (pain, fatigue, feeling of tiredness).
Psychosomatic assessment | Baseline and up to three weeks
  The Brief Symptom Checklist (LSB-50) will be used. It is a clinical instrument for the identification and assessment of psychological and psychosomatic symptoms in adults. It has been developed from the authors' experience with other symptom measurement questionnaires.
  The questionnaire is composed of 7 main scales (Obsessive Sensitivity, Anxiety, Hostility, Somatisation, Depression, Strict Sleep and Extended Sleep); 2 subscales (Sensitivity and Obsessive-Compulsion) and 1 Psychopathological Risk scale. It allows 3 global indices to be obtained (Global Severity Index, Number of Positive Symptoms and Positive Symptom Intensity Index), each of which is indicative of different aspects of general psychopathological distress.
Sleep assessment (time elapsed between each sleep phase) | Baseline and up to three weeks
  Using the polysomnography technique, the duration of the different phases of sleep will be evaluated.
  Polysomnography is a non-invasive and painless test that allows the study of sleep, its phases (REM and non-REM) and also its various alterations. In order to recognise which phase of sleep the patient is in, and to quantify the time that elapses during the phase, polysomnography simultaneously performs an electroencephalogram (EEG), detects muscle activity with a surface electromyogram, usually submental (EMG), eye movements with an electrooculogram (EOG) and body position using sensors on the limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Gómez Garrido, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Hugo Gómez Garrido, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bradley LA. Pathophysiology of fibromyalgia. Am J Med. 2009 Dec;122(12 Suppl):S22-30. doi: 10.1016/j.amjmed.2009.09.008. PMID 19962493
- [Result] Dadabhoy D, Crofford LJ, Spaeth M, Russell IJ, Clauw DJ. Biology and therapy of fibromyalgia. Evidence-based biomarkers for fibromyalgia syndrome. Arthritis Res Ther. 2008;10(4):211. doi: 10.1186/ar2443. Epub 2008 Aug 8. PMID 18768089
- [Result] Hauser W, Ablin J, Fitzcharles MA, Littlejohn G, Luciano JV, Usui C, Walitt B. Fibromyalgia. Nat Rev Dis Primers. 2015 Aug 13;1:15022. doi: 10.1038/nrdp.2015.22. PMID 27189527
- [Result] Yunus MB. Fibromyalgia and overlapping disorders: the unifying concept of central sensitivity syndromes. Semin Arthritis Rheum. 2007 Jun;36(6):339-56. doi: 10.1016/j.semarthrit.2006.12.009. Epub 2007 Mar 13. PMID 17350675